CLINICAL TRIAL: NCT05082623
Title: The Effect of Music on Delirium, Pain, Need of Sedation, Anxiety and Vital Parameters in Patients Receiving Ventilator Support in Intensive Care
Brief Title: The Effect of Music on Delirium, Pain, Need of Sedation, Anxiety and Vital Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Öznur ERBAY DALLI, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Music in intensive care
Record Dates: First submitted 2021-09-20; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Delirium; Pain; Sedation; Anxiety; Music; Intensive Care Unit Delirium
Keywords: delirium; intensive care; music
MeSH Terms: conditions — Delirium; Pain; Anxiety Disorders | interventions — Music Therapy; Ear Protective Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): "MusiCure®" compositions specially composed for the music group will be performed twice a day, between 10.00-11.00 a.m. and 14.00-15.00 p.m., for five days with headphones and a music player. Before the application, the sound level of the ICU environment will be measured with a decibel meter. At the 0th minute of the music application, at the 30th minute after starting the music, and at the 60th minute after the end of the music, the characteristics of delirium, pain, sedation level, anxiety and vital parameters will be recorded with data collection tools.
  Interventions: Other: Music
- Earplug group (Active Comparator): In this group, patients will be given only earplugs. Before the application, the sound level of the ICU environment will be measured with a decibel meter. At the 0th minute of the intervention, at the 30th minute after starting intervention, and at the 60th minute after the end of the intervention, the characteristics of delirium, pain, sedation level, anxiety and vital parameters will be recorded with data collection tools.
  Interventions: Other: Earplug
- Control group (No Intervention): The control group involves neither music intervention nor using earplug.

INTERVENTIONS:
Other: Music — Music medicine
  Arms: Music group
Other: Earplug — Earplug with noise cancelling
  Arms: Earplug group

SUMMARY:
The purpose of this study is to test the effect of a twice daily, 60-minute, nurse initiated, music listening intervention on patients followed in the ICU with MV support as compared to patients who receive care as usual and ear plugs.

DETAILED DESCRIPTION:
Delirium is an acute disorder of consciousness and cognitive function that occurs frequently in critical care settings. Many critically ill patients (e.g., up to 80% of patients) experience ICU delirium due to underlying medical or surgical health problems, recent surgical or other invasive procedures, medications, or various noxious stimuli (e.g., underlying psychological stressors, mechanical ventilation [MV], noise, light, patient care interactions, and drug-induced sleep disruption or deprivation). Delirium contributes to adverse outcomes such as increased mortality and morbidity, longer length of ICU stays, prolonged MV, costlier hospitalizations, and cognitive impairment after hospital discharge. The Society of Critical Care Medicine (SCMM) Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU (PADIS) recommend non-pharmacological interventions of preventing delirium and other symptoms. Music, which is one of the non-pharmacological applications, is one of the cognitive-behavioral treatment methods applied in the field of ICU as in many other fields. Music is easy method to apply and has no side effects and contributes to physical, psychological, emotional and spiritual healing. In the literature, it is seen that music intervention studies applied to patients followed in the ICU mostly focus on the effects on anxiety, pain, non-invasive ventilation tolerance, and stress response (heart rate, blood pressure, respiratory rate). The relationship between intensive care delirium and all these symptoms (pain, agitation, anxiety, stress response, etc.) and their interaction with each other have been clarified in the light of evidence-based guidelines and studies. Therefore, the aim of this study is to examine the effects of music applied to patients followed in the ICU with MV support on delirium, pain, need for sedation, anxiety and vital parameters.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years,
* Admitted to the ICU as of the start of the study and planned to be followed up in the ICU for at least 24 hours,
* Needing invasive MV for at least 24 hours,
* Pre-deliric score > 20%
* At least one positive delirium according to CAM-ICU,
* GCS score > 8,
* RASS score ≥ -3,
* Hemodynamically stable,
* CPOT score ≥ 3

Exclusion Criteria:

* Hearing or vision problems,
* Diagnosed with psychiatric illness,
* Diagnosed with dementia,
* Having acute neurological injury,
* Alcohol/drug poisoning
* Hemodynamically unstable and treated with high-dose inotropic/vasopressor medication,
* Pregnant,
* Planned to be followed in ICU for less than 24 hours,
* Does not need MV,
* GCS score ≤ 8,
* RASS score < -3,
* Patients referred from another ICU

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Delirium | Date of study enrollment through 12 months.
  The delirium event assessed twice daily by trained research nurse using the CAM-ICU. The diagnosis of delirium is based on the presence of two major criteria (i.e. acute or fluctuating onset plus lack of attention) and at least one of the minor criteria (disorganized thinking or altered consciousness level).

SECONDARY OUTCOMES:
Delirium severity | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  In case of positive delirium, its severity assessed twice daily by trained research nurse using the CAM-ICU-7. CAM-ICU-7 is a seven point scale (0-7), derived from the RASS and the CAM-ICU.
Pain severity | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Pain assessed by trained research nurse utilizing the Critical Care Pain Observation Tool (CPOT) a valid and reliable instrument in critically ill patients with and without delirium. The CPOT has 4 components: facial expression, body movements, muscle tension, and compliance with the ventilator for intubated patients or vocalization for extubated patients. Each component is scored from 0 to 2 with a possible total score ranging from 0 to 8. A CPOT ≥ 3 is indicative of significant pain.
Need of sedation | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Sedation level assessed by trained research nurse using the Richmond Agitation-Sedation Scale (RASS). It is a ranking scale with 10-level (+4 "combative" to -5 "unarousable") used to measure the agitation or sedation level of a person.
Anxiety level | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Anxiety level assessed by trained research nurse using Face Anxiety Scale. The scale is composed of five face types. The face type in the left-hand corner indicates an absence of anxiety, while anxiety increases towards the faces in the right-hand corner. When patient scores were three or above, their anxiety was determined to be medium to high.
Systolic/diastolic blood pressure | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Changes in the systolic/diastolic blood pressure (mm/Hg). Blood pressure was recorded from monitor of patient.
Heart rate | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Changes in the heart rate. Heart rate was measured as number of heartbeats in a per minute from monitor of patient.
Respiratory rate | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Changes in the respiratory rate. Respiratory rate was measured as number of breaths in a per minute from monitor of patient.
Oxygen saturation | 2 times daily, before, midst and after each intervention for up to 5 days while in the ICU post randomization
  Changes in the oxygen saturation. Saturation was recorded from monitor of patient.

OTHER OUTCOMES:
Length of ICU stay | During ICU stay (from randomization until ICU discharge, or death, or 1 year follow-up)
  The total days of ICU stay.
Duration of mechanical ventilation | During ICU stay (from randomization until ICU discharge, or death, or 1 year follow-up)
  The total days of mechanical ventilation.
Delirium duration | During ICU stay (from randomization until ICU discharge, or death, or 1 year follow-up)
  The delirium duration will be calculated when the patient is first considered to have delirium to the last time that patient is not supposed to have delirium based on CAM-ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided